CLINICAL TRIAL: NCT00511862
Title: TheraSphere for the Treatment of Liver Metastases: An Open Label Trial of TheraSphere in Patients With Liver Metastases From Primary Colorectal Cancer, Neuroendocrine Cancer or Non-colorectal/Non-neuroendocrine Cancer
Brief Title: TheraSphere for the Treatment of Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G040148
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer; Carcinoma, Neuroendocrine; Neoplasm Metastasis
Keywords: TheraSphere; radioactive microspheres; Yttrium-90; Yttrium glass microspheres
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Neuroendocrine; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TheraSphere (Experimental): Single arm, TheraSphere Yttrium 90 glass microspheres at 120 Gy +/- 10%; stratified by type of disease (colorectal cancer, neuroendocrine cancer, non-colorectal/non-neuroendocrine cancer
  Interventions: Device: Yttrium 90 glass microspheres

INTERVENTIONS:
Device: Yttrium 90 glass microspheres — 120 Gy unilobar or bilobar infusion with the second infusion occurring 3-7 weeks following treatment of the first lobe
  Other Names: TheraSphere

SUMMARY:
This study will evaluate Liver Progression Free Survival (PFS) and safety of TheraSphere treatment at doses of 120 Gy +/1 10% in patients at least 18 years of age diagnosed with metastatic disease to the liver that cannot be treated or is progressing following treatment with systemic or other liver-directed therapies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* diagnosis of metastatic disease to the liver that is refractory to, or inappropriate for, other systemic or liver-directed therapies
* unresectable liver metastases
* target tumors measurable using standard imaging techniques
* tumor replacement < or = 50% of total liver volume (visual estimation by investigator)
* Hypervascular tumors (visual estimation by investigator)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* minimum one month since most recent prior cancer therapy with the exception of patients receiving Sandostatin for neuroendocrine cancer
* patient informed consent

Exclusion Criteria:

* At risk of hepatic or renal failure within 21 days of treatment (serum creatinine > 2.0 mg/dL unless on dialysis; serum bilirubin ≥ 2.0 mg/dL; albumin < 2.0 mg/dL or any history of hepatic encephalopathy)
* contraindications to angiography and selective visceral catheterization including any non-correctable bleeding diathesis or coagulopathy, severe peripheral vascular disease or history of non-management allergy or intolerance to contrast, narcotics, sedatives or atropine
* severe liver dysfunction or presentation of pulmonary insufficiency or clinically evident history of chronic obstructive pulmonary disease
* cirrhosis or portal hypertension
* prior external beam radiation treatment to the liver
* prior TheraSphere treatment to the liver
* any intervention for, or compromise of the Ampulla of Vater
* clinically evident ascites (trace ascites on imaging is acceptable)
* any continuing complications of prior cancer therapy that have not improved or resolved prior to 21 days before first TheraSphere treatment
* significant life-threatening extrahepatic disease in judgment of physician
* concurrent enrollment in another study
* alternative available therapies in judgement of physician
* evidence on technetium-99m macroaggregated albumin scan that shows lung shunting > 30 Gy cumulative limit
* evidence on technetium-99m macroaggregated albumin scan showing potential for deposition of microspheres to the gastrointestinal tract that cannot be eliminated by catheter placement or corrective action using standard angiographic techniques
* positive serum pregnancy test in women of childbearing potential
* co-morbid disease or condition that puts the patient at undue risk or precludes use of TheraSphere in judgment of physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al Benson III, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern Memorial Hospital, Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - John Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Albany Medical Center, Albany, New York
  - Medical College of Wisconsin, Froedtert Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 patients recruited from January 19, 2007 to October 7, 2009
Pre-assignment Details: Patients were assigned to groups on the basis of type of primary cancer - colorectal cancer; neuroendocrine cancer or non-colorectal/non-neuroendocrine. Subjects who unable to receive TheraSphere (target dose 120 Gy) due to vascular shunting to the lungs or GI tract were not enrolled in the study and did not receive yttrium 90 glass microspheres.
Groups:
- Colorectal Cancer: Colorectal cancer patients with liver metastatic disease, refractory to standard of care therapy who received intrahepatic TheraSphere yttrium-90 glass microspheres (target dose 120 Gy) on Day 0
- Neuroendocrine Cancer: Neuroendocrine cancer patients with liver metastatic disease, refractory to standard of care therapy who received intrahepatic TheraSphere yttrium-90 glass microspheres (target dose 120 Gy) on Day 0
- Non-Colorectal/Non-neuroendocrine: Patients with liver metastatic disease not arising from colorectal cancer or neuroendocrine cancer, refractory to standard of care therapy who received intrahepatic TheraSphere yttrium-90 glass microspheres (target dose 120 Gy) on Day 0
Period: Overall Study
Arm/Group | Colorectal Cancer | Neuroendocrine Cancer | Non-Colorectal/Non-neuroendocrine
Started | 61 | 43 | 47
Completed | 61 | 43 | 47
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects treated with TheraSphere were enrolled and assigned to groups based on their primary cancer type. The total population and each subgroup population was analyzed for safety, progression and survival endpoints. In the neuroendocrine group, a median overall survival was not achieved so a post-hoc analysis of 2 year survival was performed.
Groups:
- Colorectal Cancer: colorectal cancer patients with liver metastatic disease, refractory to standard of care therapy
- Neuroendocrine Cancer: neuroendocrine cancer patients with liver metastatic disease, refractory to standard of care therapy
- Non-Colorectal/Non-neuroendocrine: patients with liver metastatic disease not arising from colorectal cancer or neuroendocrine cancer, refractory to standard of care therapy
- Total: Total of all reporting groups
Arm/Group | Colorectal Cancer | Neuroendocrine Cancer | Non-Colorectal/Non-neuroendocrine | Total
Number analyzed (Participants) | 61 | 43 | 47 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 22 | 20 | 71
  >=65 years | 32 | 21 | 27 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.92) | 61.8 (13.71) | 66.1 (8.52) | 63.7 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 23 | 67
  Male | 36 | 24 | 24 | 84
Region of Enrollment [Number; unit: participants]
  United States | 61 | 43 | 47 | 151

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Progression-free Survival According to Response Evaluation Criterian in Solid Tumors (RECIST)
Description: Progression per RECIST v 1.0 is defined as at least 20% increase in the sum of the longest diameter of target lesions, taking as the reference the smallest sum of longest diameters recorded since treatment started, or unequivocal progression of existing non-target lesion or appearance of new lesions. A maximum of 5 target lesions per organ are assessed. To assess the impact of a non-systemic local therapy on progression, for the purposes of this trial, hepatic progression was defined as at least a 20% increase in the sum of the longest diameter of target hepatic lesions. Hepatic progression-free survival is the time from the day of first treatment with TheraSphere to determination of hepatic progression.
Time Frame: From the date of first treatment until date of first documented progression; median patient follow-up 30 months
Population: Patients receiving at least one TheraSphere treatment with images evaluable by RECIST
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Patients: All patients in colorectal cancer, neuroendocrine cancer and non-colorectal/non-neuroendocrine groups
Arm/Group | Colorectal Cancer | Neuroendocrine Cancer | Non-Colorectal/Non-neuroendocrine | All Patients
Number analyzed (Participants) | 58 | 43 | 46 | 147
Months | 3.0 [2.0 to 5.8] | 17.9 [13.5 to 19.5] | 2.9 [1.3 to 3.3] | 3.4 [3.0 to 6.5]

2. Secondary Outcome: Overall Survival
Description: Duration of survival from date of first TheraSphere treatment to date of death or censored to last known date alive.
Time Frame: Time from first TheraSphere treatment to death; median follow up 30 months
Population: In the neuroendocrine group, a median overall survival was not achieved so a post-hoc analysis of 2 year survival was performed in Outcome Measure 3.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Non Colorectal/Non-Neuroendocrine: Patients with metastatic liver disease arising from primary cancers other than colorectal or neuroendocrine cancer who received intrahepatic TheraSphere yttrium-90 glass microspheres (target dose 120 Gy) on Day 0
Arm/Group | Colorectal Cancer | Non Colorectal/Non-Neuroendocrine | All Patients
Number analyzed (Participants) | 61 | 47 | 151
Months | 8.8 [6.6 to 11.9] | 10.4 [6.6 to 14.6] | 13.6 [11.1 to 16.1]

3. Post Hoc Outcome: 2 Year Survival
Description: The percentage of patients in the neuroendocrine group alive at 2 years
Time Frame: 24 months from treatment
Measure: Number; unit: percentage of treated subjects
Arm/Group | Neuroendocrine Cancer
Number analyzed (Participants) | 43
percentage of treated subjects | 79.1

ADVERSE EVENTS:
Time Frame: All adverse events collected for 3 months, device-related adverse events captured to month 18
Groups:
- TheraSphere: total population receiving at least one TheraSphere treatment
Arm/Group | TheraSphere
Serious Adverse Events (participants affected / at risk) | 21/151
Other Adverse Events (participants affected / at risk) | 139/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TheraSphere (N=151)
Abdominal or epigastric pain (Nervous system disorders) | 5 (5)
Death (General disorders) | 2 (2)
Decreased platelets (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Esophagial varices (Gastrointestinal disorders) | 1 (1)
GI hemorrhage (Blood and lymphatic system disorders) | 1 (1)
GI ulcer (Gastrointestinal disorders) | 2 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Liver dysfunction/failure (Hepatobiliary disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Obstruction (Gastrointestinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Thrombosis/embolus (Vascular disorders) | 1 (1)
Vessel injury - lower extremity artery (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TheraSphere (N=151)
ALT > ULN (Metabolism and nutrition disorders) | 26 (26)
AST >ULN (Metabolism and nutrition disorders) | 36 (36)
Alkaline phosphatase >ULN (Metabolism and nutrition disorders) | 56 (56)
Anorexia (Metabolism and nutrition disorders) | 36 (36)
Bilirubin >ULN (Metabolism and nutrition disorders) | 19 (19)
Constipation (Gastrointestinal disorders) | 11 (11)
Fatigue (General disorders) | 91 (91)
Hypoalbuminemia < LLN (Metabolism and nutrition disorders) | 19 (19)
Lymphopenia (Blood and lymphatic system disorders) | 16 (16)
Nausea (Gastrointestinal disorders) | 59 (59)
Pain (Nervous system disorders) | 62 (62)
Vomitting (Gastrointestinal disorders) | 19 (19)
Weight loss (General disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No